CLINICAL TRIAL: NCT05434221
Title: Development and Evaluation of a Communication Skill Training Program for Occupational Therapy Interns
Brief Title: Communication Skill Training Program for Occupational Therapy Interns
Acronym: COPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202006114RINC
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Education, Medical
Keywords: Communication skill; occupational therapy; intern

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): interns in the experiment group receive COPE during their internship.
  Interventions: Other: COPE
- Control group (No Intervention): interns in the control group do not receive any specific communication training during their internship.

INTERVENTIONS:
Other: COPE — The experimental group receives the COPE during their internships. The COPE consists of two part: (1) communication skills teaching and simulation practice; (2) clinical communication teaching: record the clinical treatment process of the interns and turn them into verbatim drafts. Experts then complied the strengths and weaknesses of the interns' communication skills based on the verbatim manuscripts and gave feedback on the interns' communication skills.
  The interns in the experimental group will participate 1 time of the communication skills teaching and simulation practice, and 3 times of the clinical communication teaching in three months.
  Arms: Experiment group

SUMMARY:
Effective communication is one of important skills in occupational therapy (OT) practice, affecting the effectiveness and quality of therapy. Although there are only a few courses on communication skills related to OT, there is a lack of a complete, suitable, and evidence-based OT communication skills teaching programs that can effectively improve the interns' communication skills. The purpose of the study is to develop a communication skills training program for occupational therapy interns in physical dysfunction practice (COPE), and examine the effectiveness of COPE.

ELIGIBILITY:
Inclusion Criteria:

[interns]

* age ≥ 20 years
* an intern of occupational therapy

[patients]

* age ≥ 20 years
* enable to communicate with the others

Exclusion Criteria:

[interns]

* unwilling to be recorded

[patients]

* have communication barriers
* unwilling to be recorded

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Experts assessed interns' communication skills：Gap-Kalamazoo Communication Skills Assessment Forms (GKCSAF)-Faculty version | during procedure
  The experts will use the questionnaire named GKCSAF (faculty version) to assess interns' communication skills via verbatim draft of the audio-recording.
  The GKCSAF contains 9 items: build a relationship, open the discussion, gather information, understand the patients' perspective, share information, reach agreement, provide closure, demonstrate empathy, and communicate accurate information. Each item is rated on a 5-point Likert-type scale. The total score ranges from 5 to 45. The higher scores indicate better communication skills.

SECONDARY OUTCOMES:
Patients or caregivers assessed interns' communication skills：Gap-Kalamazoo Communication Skills Assessment Forms (GKCSAF)-patient/caregiver version | during procedure
  The patients will use the questionnaire named GKCSAF (patient/caregiver version) to assess the interns' communication skills after their occupation therapy.
  The items and the score range are the same with the faculty version.
Interns self-reported communication skills：Gap-Kalamazoo Communication Skills Assessment Forms (GKCSAF)-self-assessment version | during procedure
  The interns will use the GKCSAF (self-assessment version) to assess their communication skills via verbatim draft of the audio-recording after they communicate with the patients.
  The items and the score range are the same with the faculty and patient/caregiver version.
Patients' engagements in occupational therapy：Occupational Therapy Engagement Scale (OTES) | during procedure
  The experts will use OTES to assess patients' engagement in occupational therapy for one week.
  The OTES is a questionnaire which is designed to assess patients' engagement level in occupational therapy. The OTES contains 12 items, such as "commit in therapy activities without being urged", "sustain attention until the end of one therapeutic activity", and so on. Each item is rated on a 4-point scale. The total score ranges from 0 to 36. A higher sum score indicates a higher level of engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Calhoun AW, Rider EA, Peterson E, Meyer EC. Multi-rater feedback with gap analysis: an innovative means to assess communication skill and self-insight. Patient Educ Couns. 2010 Sep;80(3):321-6. doi: 10.1016/j.pec.2010.06.027. Epub 2010 Jul 17. PMID 20638814
- [Background] Peterson EB, Calhoun AW, Rider EA. The reliability of a modified Kalamazoo Consensus Statement Checklist for assessing the communication skills of multidisciplinary clinicians in the simulated environment. Patient Educ Couns. 2014 Sep;96(3):411-8. doi: 10.1016/j.pec.2014.07.013. Epub 2014 Jul 19. PMID 25103180
- [Background] Wu TY, Lien BY, Lequerica AH, Lu WS, Hsieh CL. Development and Validation of the Occupational Therapy Engagement Scale for Patients with Stroke. Occup Ther Int. 2019 Mar 6;2019:3164254. doi: 10.1155/2019/3164254. eCollection 2019. PMID 30962799